CLINICAL TRIAL: NCT04058717
Title: Randomized Trial of Low Nicotine Cigarettes Plus Electronic Cigarettes in Smokers
Brief Title: Low Nicotine Cigarettes Plus Electronic Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jonathan Foulds, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY12579; R01DA048428 (NIH)
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: 2 X 2 factorial design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NNC cigarettes + High Nicotine Containing E-cigarette (Experimental): Participants are provided with normal nicotine content (NNC) cigarettes (11.6 mg nicotine/cigarette) plus e-cigarette with high nicotine e-liquid.
  Interventions: Other: Normal Nicotine Content research cigarettes; Other: High Nicotine e-cigarette
- NNC cigarettes + Zero Nicotine Containing E-cigarette (Experimental): Participants are provided with normal nicotine content (NNC) cigarettes (11.6 mg nicotine/cigarette) plus e-cigarette with zero nicotine e-liquid.
  Interventions: Other: Normal Nicotine Content research cigarettes; Other: Zero Nicotine e-cigarette
- VLNC cigarettes + High Nicotine Containing E-cigarette (Experimental): Participants are provided with very low nicotine content (VLNC) cigarettes (0.2 mg nicotine/cigarette) plus e-cigarette with high nicotine e-liquid.
  Interventions: Other: High Nicotine e-cigarette; Other: Very Low Nicotine Content research cigarettes
- VLNC cigarettes + Zero Nicotine Containing E-cigarette (Experimental): Participants are provided with very low nicotine content (VLNC) cigarettes (0.2 mg nicotine/cigarette) plus e-cigarette with zero nicotine e-liquid
  Interventions: Other: Very Low Nicotine Content research cigarettes; Other: Zero Nicotine e-cigarette

INTERVENTIONS:
Other: Normal Nicotine Content research cigarettes — Research cigarettes with 11.6 mg nicotine/cigarette.
  Arms: NNC cigarettes + High Nicotine Containing E-cigarette; NNC cigarettes + Zero Nicotine Containing E-cigarette
Other: High Nicotine e-cigarette — E-cigarette containing high nicotine e-liquid
  Arms: NNC cigarettes + High Nicotine Containing E-cigarette; VLNC cigarettes + High Nicotine Containing E-cigarette
Other: Very Low Nicotine Content research cigarettes — Research cigarettes with 0.2 mg nicotine/cigarette.
  Arms: VLNC cigarettes + High Nicotine Containing E-cigarette; VLNC cigarettes + Zero Nicotine Containing E-cigarette
Other: Zero Nicotine e-cigarette — E-cigarette containing zero nicotine e-liquid
  Arms: NNC cigarettes + Zero Nicotine Containing E-cigarette; VLNC cigarettes + Zero Nicotine Containing E-cigarette

SUMMARY:
This study aims to determine the health effects of very low nicotine content in cigarettes, in conjunction with the availability of nicotine-containing electronic cigarettes (e-cigs) among smokers with mental health conditions (SMHC).

DETAILED DESCRIPTION:
The specific objective of this study is to recruit a cohort of 240 current exclusive daily SMHC (diagnosed using the MINI International Neuropsychiatric Interview) and to measure a comprehensive battery of behavioral and health indicators at 4, 8, 12 and 16 weeks after being randomized to use either normal nicotine content (NNC) Spectrum cigarettes (11.6 mg nicotine/cigarette) or very low nicotine content (VLNC) Spectrum cigarettes (0.2 mg nicotine/cigarette) while also having access to an electronic cigarette (containing either 0 nicotine or high nicotine e-liquid) in a randomized double-blind, placebo-controlled, 2 by 2 design. All participants will be followed up with a study visit 4 weeks after the final randomized visit to identify whether they have continued to use e-cigs/cigarettes and to assess their motivation in smoking abstinence.

Our central hypothesis is that key markers of harms to health (e.g. urinary NNAL, exhaled carbon monoxide, measures of addiction, and mental distress) will be significantly improved among SMHC who are provided VLNC cigarettes and high nicotine e-cigs.

ELIGIBILITY:
Inclusion Criteria:

* Smoke >5 cigarettes per day for at least the prior 12 months
* Smoke regular, filtered cigarettes or machine-rolled cigarettes with a filter
* Exhaled CO measurement of ≥ 6 parts per million at baseline
* No serious cigarette smoking quit attempt or use of any FDA-approved smoking cessation medication in the prior 30 days (includes any nicotine replacement, varenicline, bupropion [used specifically as a quitting aid])
* No plans to quit smoking within the next 3 weeks
* Must be willing to both switch to a different type of cigarette that may contain a different amount of nicotine and to try an e-cig to substitute for some of their cigarettes
* Must be willing and able to respond to contacts from study staff or attend visits over the study period (not planning to move, not planning extended vacation, no planned surgeries)
* 9. Must meet lifetime diagnostic criteria for a current or lifetime unipolar or bipolar mood disorder (e.g. major depressive disorder, major depressive episode, manic episode, hypomanic episode, bipolar disorder), an anxiety disorder (e.g. panic disorder, obsessive-compulsive disorder, post-traumatic stress disorder, , agoraphobia, social anxiety disorder, generalized anxiety disorder), a psychotic disorder (e.g. mood disorder or other psychotic disorder), or an eating disorder (e.g. anorexia or bulimia) based on the MINI-International Neuropsychiatric Interview Standard (MINI) (version 7.0.2)
* Able to read and write in English
* Able to understand and give informed consent
* Access to a computer/smartphone with e-mail and a reliable internet connection

Exclusion Criteria:

* Women who are pregnant and/or nursing or trying to become pregnant
* Unstable or significant medical condition in the past 3 months (e.g., recent heart attack or other serious heart condition, stroke, severe angina, high blood pressure [systolic >159 mmHg or diastolic >99 mmHg during screening)
* Respiratory diseases (e.g., exacerbations of asthma or COPD, require oxygen, require oral prednisone), kidney (e.g., dialysis) or liver disease (e.g., cirrhosis), severe immune system disorders (e.g., uncontrolled HIV/AIDS, multiple sclerosis symptoms) or any medical disorder/medication that may affect participant safety or biomarker data
* Uncontrolled mental illness or substance abuse, or inpatient treatment for these in the past 6 months
* Current suicide risk on clinical assessment (above "low risk" score (or ≥ 9) on MINI diagnostic interview suicide module during screening (34))
* Use of any non-cigarette nicotine delivery product (e.g., pipe, cigar, dip, chew, snus, hookah, e-cig, strips or sticks, IQOS) in the past 7 days at screening
* Use of an e-cig for 5 or more days in the past 28 days or any use in the past 7 days at screening
* Use of marijuana or other illegal drugs/prescription drugs for non-medical use daily/almost daily or weekly in the past 3 months per NIDA Quick Screen
* Any known allergy to propylene glycol or vegetable glycerin
* Surgery requiring general anesthesia in the past 6 weeks
* Unwilling to remain on one flavor of cigarette (regular or menthol) for the duration of the trial
* Previous use of SPECTRUM research cigarettes in the past 6 months
* Other member of household currently participating in the study
* History of a seizure disorder or had a seizure in the past 12 months
* Currently taking or have taken medications prescribed to prevent seizures (such as Carbamazepine or Phenobarbital). Using seizure medications for off-label use (indications other than treatment for seizures) will not be included as an exclusion, these will be assessed on a case-by-case basis

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Foulds, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 88 participants consented and enrolled in the pre-randomization phase of the study. Eight participants were lost to follow-up or withdrawn from the study before being randomized to a study intervention. Therefore, 80 participants were randomized to a study intervention.
Period: Randomization Period
Arm/Group | NNC Cigarettes + High Nicotine Containing E-cigarette | NNC Cigarettes + Zero Nicotine Containing E-cigarette | VLNC Cigarettes + High Nicotine Containing E-cigarette | VLNC Cigarettes + Zero Nicotine Containing E-cigarette
Started | 20 | 20 | 20 | 20
Completed | 17 | 13 | 13 | 13
Not Completed | 3 | 7 | 7 | 7
Not completed — Lost to Follow-up | 2 | 3 | 4 | 4
Not completed — Withdrawal by Subject | 1 | 3 | 3 | 3
Not completed — PI decision | 0 | 1 | 0 | 0
Period: Week 20 Follow up
Arm/Group | NNC Cigarettes + High Nicotine Containing E-cigarette | NNC Cigarettes + Zero Nicotine Containing E-cigarette | VLNC Cigarettes + High Nicotine Containing E-cigarette | VLNC Cigarettes + Zero Nicotine Containing E-cigarette
Started | 17 | 13 | 13 | 13
Completed | 15 | 13 | 13 | 11
Not Completed | 2 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NNC Cigarettes + High Nicotine Containing E-cigarette | NNC Cigarettes + Zero Nicotine Containing E-cigarette | VLNC Cigarettes + High Nicotine Containing E-cigarette | VLNC Cigarettes + Zero Nicotine Containing E-cigarette | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (9.2) | 51.2 (10.4) | 44.6 (9) | 47.8 (12.1) | 46.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 12 | 18 | 12 | 60
  Male | 2 | 8 | 2 | 8 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 2 | 7
  White | 18 | 17 | 18 | 18 | 71
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 20 | 80
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 22 (11.7) | 18.8 (9.9) | 22.4 (8.6) | 17.6 (9.8) | 20.2 (10.1)

OUTCOME MEASURES:

1. Primary Outcome: Urinary NNAL (4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol)
Description: Measure of tobacco-specific nitrosamine
Time Frame: Week 16
Population: The Overall Number of Participants Analyzed includes participants with non-missing values at Week 16. Therefore, in one of the groups, 20 people were randomized and 13 people completed the randomization phase, but only 12 of the samples could be analyzed.
Measure: Mean (Standard Deviation); unit: pg/mg creatinine
Arm/Group | NNC Cigarettes + High Nicotine Containing E-cigarette | NNC Cigarettes + Zero Nicotine Containing E-cigarette | VLNC Cigarettes + High Nicotine Containing E-cigarette | VLNC Cigarettes + Zero Nicotine Containing E-cigarette
Number analyzed (Participants) | 17 | 13 | 12 | 13
pg/mg creatinine | 505.6 (432.7) | 459.1 (312.8) | 373.3 (553.1) | 180.5 (218.2)
Statistical Analysis 1: Comparison: NNC Cigarettes + High Nicotine Containing E-cigarette vs NNC Cigarettes + Zero Nicotine Containing E-cigarette vs VLNC Cigarettes + High Nicotine Containing E-cigarette vs VLNC Cigarettes + Zero Nicotine Containing E-cigarette; Test type: Other; p = 0.017, Kruskal-Wallis; H-statistic = 10.23

2. Secondary Outcome: Exhaled Carbon Monoxide
Description: Measure of cigarette smoke exposure
Time Frame: Week 16
Population: The Overall Number of Participants Analyzed includes participants with non-missing values at Week 16. In two of the groups, 1 person had missing CO values.
Measure: Mean (Standard Deviation); unit: parts per million
Arm/Group | NNC Cigarettes + High Nicotine Containing E-cigarette | NNC Cigarettes + Zero Nicotine Containing E-cigarette | VLNC Cigarettes + High Nicotine Containing E-cigarette | VLNC Cigarettes + Zero Nicotine Containing E-cigarette
Number analyzed (Participants) | 17 | 12 | 12 | 13
parts per million | 23.6 (9.4) | 25.2 (14.6) | 21.9 (24.5) | 12.6 (10.3)
Statistical Analysis 1: Comparison: NNC Cigarettes + High Nicotine Containing E-cigarette vs NNC Cigarettes + Zero Nicotine Containing E-cigarette vs VLNC Cigarettes + High Nicotine Containing E-cigarette vs VLNC Cigarettes + Zero Nicotine Containing E-cigarette; Test type: Other; p = 0.056, Kruskal-Wallis; H-statistic = 7.57

3. Secondary Outcome: Kessler-6 Score
Description: Measure of serious psychological distress. This scale is a brief, self-report tool used to assess psychological distress. Scores range from 0-24, with higher scores indicating greater distress
Time Frame: Week 16
Population: The Overall Number of Participants Analyzed includes all participants with non-missing values at Week 16. In the VLNC cigarettes + High Nicotine Containing E-cigarette group, two participants did not complete the entire Week 16 visit, but they did complete the Kessler-6 survey for Week 16. Therefore, their Kessler-6 survey data are included in this analysis even though they were not included in the final sample size for Week 16, resulting in a sample size of n=15 for this group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNC Cigarettes + High Nicotine Containing E-cigarette | NNC Cigarettes + Zero Nicotine Containing E-cigarette | VLNC Cigarettes + High Nicotine Containing E-cigarette | VLNC Cigarettes + Zero Nicotine Containing E-cigarette
Number analyzed (Participants) | 17 | 13 | 15 | 13
score on a scale | 6.9 (5.9) | 5.7 (5.1) | 5.4 (5.9) | 5.9 (4.3)
Statistical Analysis 1: Comparison: NNC Cigarettes + High Nicotine Containing E-cigarette vs NNC Cigarettes + Zero Nicotine Containing E-cigarette vs VLNC Cigarettes + High Nicotine Containing E-cigarette vs VLNC Cigarettes + Zero Nicotine Containing E-cigarette; Test type: Other; p = 0.74, Kruskal-Wallis; H-statistic = 1.26

4. Secondary Outcome: Penn State Cigarette Dependence Index
Description: Measure of cigarette dependence. This 10-item scale (with scores ranging from 0 to 20) was developed to measure cigarette dependence, where a score of 0 indicates no cigarette dependence and 20 indicates maximum cigarette dependence.
Time Frame: Week 16
Population: The Overall Number of Participants Analyzed includes everyone with non-missing values at Week 16. In the VLNC cig+High Nic E-cig group, 1 person did not complete the entire Week 16 visit, but they did complete the Cig Dep survey for Week 16. Therefore, their Cig Dep survey data are included in this analysis, even though they were not included in the final sample size for Week 16, resulting in a sample size of n=14 for this group. 1 person had missing data in the VLNC cig+Zero Nic E-cig.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNC Cigarettes + High Nicotine Containing E-cigarette | NNC Cigarettes + Zero Nicotine Containing E-cigarette | VLNC Cigarettes + High Nicotine Containing E-cigarette | VLNC Cigarettes + Zero Nicotine Containing E-cigarette
Number analyzed (Participants) | 17 | 13 | 14 | 12
score on a scale | 11.9 (3) | 11.5 (2.9) | 11.8 (4.3) | 9.4 (3.2)
Statistical Analysis 1: Comparison: NNC Cigarettes + High Nicotine Containing E-cigarette vs NNC Cigarettes + Zero Nicotine Containing E-cigarette vs VLNC Cigarettes + High Nicotine Containing E-cigarette vs VLNC Cigarettes + Zero Nicotine Containing E-cigarette; Test type: Other; p = 0.248, Kruskal-Wallis; Slope = 4.13

5. Secondary Outcome: Penn State Electronic Cigarette Dependence Index
Description: Measure of e-cigarette dependence. This 10-item scale (with scores ranging from 0 to 20) was developed to measure e-cigarette dependence, where a score of 0 indicates no cigarette dependence and 20 indicates maximum e-cigarette dependence.
Time Frame: Week 16
Population: The Overall Number of Participants Analyzed includes everyone with non-missing values at Week 16. In the VLNC cig+High Nic E-cig group, 1 person did not complete the entire Week 16 visit, but they did complete the E-cig Dep survey for Week 16. Therefore, their E-cig Dep survey data are included in this analysis, even though they were not included in the final sample size for Week 16, resulting in a sample size of n=14 for this group. 2 people had missing data in the VLNC cig+0 Nic E-cig group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NNC Cigarettes + High Nicotine Containing E-cigarette | NNC Cigarettes + Zero Nicotine Containing E-cigarette | VLNC Cigarettes + High Nicotine Containing E-cigarette | VLNC Cigarettes + Zero Nicotine Containing E-cigarette
Number analyzed (Participants) | 17 | 13 | 14 | 11
score on a scale | 3.1 (3) | 5.8 (3.8) | 8.1 (5.2) | 5.8 (4.1)
Statistical Analysis 1: Comparison: NNC Cigarettes + High Nicotine Containing E-cigarette vs NNC Cigarettes + Zero Nicotine Containing E-cigarette vs VLNC Cigarettes + High Nicotine Containing E-cigarette vs VLNC Cigarettes + Zero Nicotine Containing E-cigarette; Test type: Other; p = 0.025, Kruskal-Wallis; H-statistic = 9.33

6. Secondary Outcome: Cigarette Abstinence
Description: No cigarette use in the past 7 days and exhaled carbon monoxide < 6ppm
Time Frame: Week 20
Population: This is an intent-to-treat analysis so everyone who was randomized was included in the sample analyzed, regardless of whether they completed the Week 20 assessment. Those who did not complete the Week 20 assessment were assumed to be non-abstainers. This is normal practice in smoking cessation research.
Measure: Count of Participants; unit: Participants
Arm/Group | NNC Cigarettes + High Nicotine Containing E-cigarette | NNC Cigarettes + Zero Nicotine Containing E-cigarette | VLNC Cigarettes + High Nicotine Containing E-cigarette | VLNC Cigarettes + Zero Nicotine Containing E-cigarette
Number analyzed (Participants) | 20 | 20 | 20 | 20
Participants | 1 | 1 | 4 | 4
Statistical Analysis 1: Comparison: NNC Cigarettes + High Nicotine Containing E-cigarette vs NNC Cigarettes + Zero Nicotine Containing E-cigarette vs VLNC Cigarettes + High Nicotine Containing E-cigarette vs VLNC Cigarettes + Zero Nicotine Containing E-cigarette; Test type: Other; p = 0.289, Fisher Exact

ADVERSE EVENTS:
Time Frame: 20 weeks
Description: Adverse events (AEs) were systematically collected at each study visit by asking participants about any changes in their medication, their physical or mental health, or if they needed to seek immediate medical care at an emergency room or hospital.
Arm/Group | NNC Cigarettes + High Nicotine Containing E-cigarette | NNC Cigarettes + Zero Nicotine Containing E-cigarette | VLNC Cigarettes + High Nicotine Containing E-cigarette | VLNC Cigarettes + Zero Nicotine Containing E-cigarette
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 4/20 | 4/20 | 2/20 | 1/20
Other Adverse Events (participants affected / at risk) | 7/20 | 11/20 | 6/20 | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NNC Cigarettes + High Nicotine Containing E-cigarette (N=20) | NNC Cigarettes + Zero Nicotine Containing E-cigarette (N=20) | VLNC Cigarettes + High Nicotine Containing E-cigarette (N=20) | VLNC Cigarettes + Zero Nicotine Containing E-cigarette (N=20)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pregnancy loss (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Self-injurious ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgical and Medical Procedures, other back electrodes (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NNC Cigarettes + High Nicotine Containing E-cigarette (N=20) | NNC Cigarettes + Zero Nicotine Containing E-cigarette (N=20) | VLNC Cigarettes + High Nicotine Containing E-cigarette (N=20) | VLNC Cigarettes + Zero Nicotine Containing E-cigarette (N=20)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 3 (3)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 5 (5) | 4 (4) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT04058717/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT04058717/ICF_001.pdf